CLINICAL TRIAL: NCT00002574
Title: PHASE II STUDY OF SIMULTANEOUS HOMOHARRINGTONINE (NSC 141633) AND ALPHA INTERFERON (IFN-A) THERAPY IN CHRONIC MYELOGENOUS LEUKEMIA (CML)
Brief Title: Homoharringtonine and Interferon Alfa in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02233; MDA-DM-93151; NCI-T93-0191D; CDR0000063647 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-10 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2001-10

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Interferon-alpha; Homoharringtonine

ARMS (1):
- Arm I (Experimental): Single-Agent Chemotherapy plus Biological Response Modifier Therapy. Homoharringtonine, HH, NSC-141633; plus Interferon alfa (Schering), IFN-A, NSC-377523.
  Interventions: Biological: recombinant interferon alfa; Drug: omacetaxine mepesuccinate

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: omacetaxine mepesuccinate

SUMMARY:
Phase II trial to study the effectiveness of homoharringtonine and interferon alfa in treating patients with chronic myelogenous leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy with interferon alfa may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of homoharringtonine administered simultaneously with interferon alpha in achieving complete cytogenetic response in patients with chronic myelogenous leukemia in chronic phase.

OUTLINE:

Single-Agent Chemotherapy plus Biological Response Modifier Therapy. Homoharringtonine, HH, NSC-141633; plus Interferon alfa (Schering), IFN-A, NSC-377523.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Chronic myelogenous leukemia (CML) in chronic phase
* Clonal evolution (i.e., the presence of clones other than the Ph chromosome) allowed Ph chromosome variants or complex Ph chromosome translocations are not considered disease acceleration
* Ineligible for known therapy of higher efficacy or priority
* Allogeneic bone marrow transplantation should be considered priority therapy for CML patients with a matched related donor
* No blastic phase CML (30% or more blasts in peripheral blood or bone marrow)
* No accelerated phase CML, defined as any of the following: 15% or more peripheral or marrow blasts or 30% or more blasts and promyelocytes 20% or more peripheral or marrow basophils
* Thrombocytopenia (platelets less than 100,000) unrelated to therapy
* Documented extramedullary disease outside of liver or spleen

PATIENT CHARACTERISTICS:

* Age: 15 and over
* Performance status: Zubrod 0-2
* Life expectancy: Sufficient to fully evaluate the effects of 2 courses of therapy
* Bilirubin no greater than 2.0 mg/dL
* SGOT less than 300
* Creatinine less than 2.0 mg/dL OR creatinine clearance at least 60 mL/min
* No severe heart disease (class III/IV)
* No pregnant or nursing women
* Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY:

* No prior interferon alpha
* At least 2 weeks since antileukemic therapy, with recovery required
* Patients who received hydroxyurea within the past 2 weeks and have WBC greater than 50,000 may enter protocol after discussion with the primary investigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 1994-09; Primary Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. O'Brien, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas - MD Anderson Cancer Center, Houston, Texas